CLINICAL TRIAL: NCT05868551
Title: Onchocerciasis-Associated Epilepsy, an Explorative Case-control Study With Viral Metagenomic Analysis of Onchocerca Volvulus.
Brief Title: Onchocerciasis-Associated Epilepsy, an Explorative Case-control Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Amref Health Africa (Other)
Responsible Party: Principal Investigator, Robert Colebunders, Emeritus professor, head NSETHIO research group, Global Health institute, Universiteit Antwerpen
Other Study IDs: AID 011898
Record Dates: First submitted 2023-05-08; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Onchocercal Subcutaneous Nodule; Epilepsy; Virus
Keywords: Onchocerciasis; Epilepsy; metagenomics; South Sudan; Pathogenesis
MeSH Terms: conditions — Epilepsy; Virus Diseases; Onchocerciasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — skin snips O.volvulus worms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with onchocerciasis nodules with OAE and without epilepsy: nodulectomy to extract adult worms
  Interventions: Procedure: nodulectomy

INTERVENTIONS:
Procedure: nodulectomy — incision in an onchocerciasis nodule to extract adult worms

SUMMARY:
This is an exploratory case control study with the aim to compare the Onchocerca volvulus virome between persons with onchocerciasis-associated epilepsy (OAE) and persons with onchocerciasis but without epilepsy.

The main question we want to address is: Is there a virus contained in the O. volulus worm that may have a pathogenic role in causing OAE.

In Maridi County, South Sudan, 20 persons with OAE with onchocerciasis nodules, and 20 age- and village-matched controls without OAE will be enrolled in a nodulectomy study.The adult O. volvulus worms will be extracted from the nodules and a viral metagenomic study of the worms. The O. volvulus virome of persons with and without OAE will be compared.

DETAILED DESCRIPTION:
A high prevalence of onchocerciasis-associated epilepsy (OAE) has been observed in onchocerciasis-endemic areas with high ongoing Onchocerca volvulus transmission. However, the pathogenesis of OAE remains to be elucidated. We hypothesise that the O. volvulus virome could be involved in inducing epilepsy. With this study, we aim to describe the O. volvulus virome and identify possible viruses linked to OAE.

In Maridi County, South Sudan, 20 persons with OAE with onchocerciasis nodules, and 20 age- and village-matched controls without OAE will be enrolled in the study. For each study participant, two skin snips at the iliac crest will be obtained to collect O. volvulus microfilaria, and one nodulectomy will be performed to obtain adult worms. A viral metagenomic study will be conducted on microfilariae and adult worms, and the O. volvulus virome of persons with and without OAE will be compared. Moreover, the prevalence, numbers and localisation of onchocerciasis nodules in persons with and without OAE in villages with a high prevalence of epilepsy in Maridi will be described.

ELIGIBILITY:
Inclusion Criteria:

* Onchocerciasis nodules
* Age 12-35 years old
* informed consent signed
* Living in Maridi County, Western Equatorial State, South Sudan

Exclusion Criteria:

* below the age of 12

Ages: 12 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Cases: persons with onchocerciasis nodules and OAE Controls: persons with onchocerciasis nodules without epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The O. volvulus virome of persons with onchocerciasis-associated epilepsy (OAE) and of persons with onchocerciasis but without epilepsy | 1 day
  The type of virusses present in the O. volvulus worm present in the nodules of persons with OAE and in nodules of persons without epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Colebunders, MD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Amref Health Africa, Juba, Central, South Sudan

IPD SHARING:
Plan to Share IPD: Undecided
After de-identification (text, tables, figures, and appendices), all individual participant data underlying the results reported in this article will be made available immediately and indefinitely via the Zenodo repository following publication for anyone who wishes to access the data for any purpose.

REFERENCES:
- [Derived] Hadermann A, Jada SR, Sebit WJ, Deng T, Bol YY, Siewe Fodjo JN, De Coninck L, Matthijnssens J, Mertens I, Polman K, Colebunders R. Onchocerciasis-associated epilepsy: an explorative case-control study with viral metagenomic analyses on Onchocerca volvulus. F1000Res. 2023 Dec 11;12:1262. doi: 10.12688/f1000research.138774.2. eCollection 2023. PMID 38439783